CLINICAL TRIAL: NCT03759275
Title: Perioperative Pain Management With Multi-discipline Team(pMDT) in Thoracic Surgery: a Multi-center，Prospective, Observational Study--------For the Baseline Investigation and Technical Preparation Stage
Brief Title: pMDT in Thoracic Surgery--------For the Baseline Investigation and Technical Preparation Stage
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Anhui Provincial Hospital (Other Government); Southwest Hospital, China (Other); Fujian Provincial Hospital (Other); Hebei Tumor Hospital (Other); Qianfoshan Hospital (Other); General Hospital of Shenyang Military Region (Other); Shanghai Chest Hospital (Other); Zhejiang University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Nanchang University (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); LanZhou University (Other); Lanzhou University Second Hospital (Other); Kunming General Hospital of PLA (Unknown); Renmin Hospital of Wuhan University (Other); Henan Provincial People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); The People's Hospital of Gaozhou (Other); Shanxi Provincial People's Hospital (Other Government); Liaoning Cancer Hospital & Institute (Other); First Affiliated Hospital of Chongqing Medical University (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Director of department of anesthesiology and pain management, Peking University People's Hospital
Other Study IDs: 2018PHB053-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
Keywords: pMDT; Pain; Thoracic surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage 1: For the Baseline Investigation and Technical Preparation Stage
  Interventions: Other: pMDT(Baseline Investigation)

INTERVENTIONS:
Other: pMDT(Baseline Investigation) — The pMDT(Baseline Investigation) takes multi-model analgesia as the main technical means. Multimodal perioperative analgesia refers to the combination of analgesics, adjuvant drugs and analgesic techniques with different effects throughout the perioperative period to achieve the best curative effect of reducing postoperative acute and chronic pain.

SUMMARY:
The risk of acute and chronic pain after thoracic surgery is high. The multi-disciplinary postoperative pain management strategy is the best way to control postoperative pain in thoracic surgery. Through nearly one year of experience in implementation of the pMDT in the thoracic surgery department of Peking University People's Hospital, the investigators have summarized the experience in multidisciplinary pain management and promoted this study in multi-centers across the country, hoping that this study can improve the current situation of acute pain management in patients after thoracic surgery, and at the same time, the deficiencies of this clinical protocol can be found out and improved.

DETAILED DESCRIPTION:
The postoperative acute pain refers to the acute pain (usually lasting less than 7 days) that occurs immediately after surgery, and its nature is traumatic pain. It may develop into a chronic pain, such as a neuropathic pain or a mixed pain, if it is not fully controlled at the initial state. It will seriously impact the physiology and psychology of a patient. According to the study, the postoperative acute pain is one of the risks for postoperative complications, and it may result in the death of a patient. However, the alleviation of a postoperative acute pain can shorten the duration of stay in hospital, and reduce the overall cost for treatment of a patient.

The risk of acute and chronic pain after thoracic surgery is high. The multi-disciplinary postoperative pain management strategy is the best way to control postoperative pain in thoracic surgery. Through nearly one year of experience in implementation of the pMDT in the thoracic surgery department of Peking University People's Hospital, the investigators have summarized the experience in multidisciplinary pain management and promoted this study in multi-centers across the country, hoping that this study can improve the current situation of acute pain management in patients after thoracic surgery, and at the same time, the deficiencies of this clinical protocol can be found out and improved.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75, ASA I-II;
* Patients undergoing thoracoscopic surgery;
* Patients who can understand and fill in the self-evaluation;
* Patients who signed the Informed Consent Form.

Exclusion Criteria:

* Pregnant women;
* Patients with preoperative chronic pain and long-term opioid use;
* Patients with advanced tumors who have received preoperative chemotherapy or who are expected to receive postoperative chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic surgery in Peking University People's Hospital and other multi-centers.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of postoperative pain | Up to 90 days after surgery.
  The percentage of patients with NRS score greater than 3
The degree of patients' satisfaction | 3 days after surgery.
  The degree of patients' satisfaction on pain managements. Patients were asked to give a score from 0-10 (0 means dissatisfied, 10 means very satisfied).

SECONDARY OUTCOMES:
Postoperative duration of stay in hospital | Up to 90 days after surgery.
  The duration when patients stay in hospital after surgery.
Rehospitalization rate | Up to 90 days after surgery.
  The percentage of patients who are rehospitalized.
Postoperative complication incidence rate | Up to 90 days after surgery.
  The percentage of patients with complications after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yi, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bugada D, Lavand'homme P, Ambrosoli AL, Klersy C, Braschi A, Fanelli G, Saccani Jotti GM, Allegri M; SIMPAR group. Effect of postoperative analgesia on acute and persistent postherniotomy pain: a randomized study. J Clin Anesth. 2015 Dec;27(8):658-64. doi: 10.1016/j.jclinane.2015.06.008. Epub 2015 Aug 30. PMID 26329661
- [Background] Kelley BP, Shauver MJ, Chung KC. Management of Acute Postoperative Pain in Hand Surgery: A Systematic Review. J Hand Surg Am. 2015 Aug;40(8):1610-9, 1619.e1. doi: 10.1016/j.jhsa.2015.05.024. PMID 26213198
- [Background] Lesin M, Domazet Bugarin J, Puljak L. Factors associated with postoperative pain and analgesic consumption in ophthalmic surgery: a systematic review. Surv Ophthalmol. 2015 May-Jun;60(3):196-203. doi: 10.1016/j.survophthal.2014.10.003. Epub 2014 Nov 5. PMID 25890623
- [Background] Sharp HT. Management of Postoperative Abdominal Wall Pain. Clin Obstet Gynecol. 2015 Dec;58(4):798-804. doi: 10.1097/GRF.0000000000000152. PMID 26512441
- [Background] Pogatzki-Zahn E, Kutschar P, Nestler N, Osterbrink J. A Prospective Multicentre Study to Improve Postoperative Pain: Identification of Potentialities and Problems. PLoS One. 2015 Nov 24;10(11):e0143508. doi: 10.1371/journal.pone.0143508. eCollection 2015. PMID 26600464
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Yun XD, Yin XL, Jiang J, Teng YJ, Dong HT, An LP, Xia YY. Local infiltration analgesia versus femoral nerve block in total knee arthroplasty: a meta-analysis. Orthop Traumatol Surg Res. 2015 Sep;101(5):565-9. doi: 10.1016/j.otsr.2015.03.015. Epub 2015 May 16. PMID 25987449